CLINICAL TRIAL: NCT03363438
Title: Knowledge Attitudes Behaviours and Practices Regarding HIV of Sex Workers in the French Antilles
Acronym: INTERREG SW
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: INTERREG Sex Workers
Record Dates: First submitted 2017-11-24; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- martinique
  Interventions: Other: no intervention survey
- guadeloupe
  Interventions: Other: no intervention survey

INTERVENTIONS:
Other: no intervention survey — there was no intervention this was a survey

SUMMARY:
The aim of the study was to determine the knowledge attitudes, behaviours and practices of sex workers regarding HIV in Martinique, guadeloupe and Saint martin.

ELIGIBILITY:
Inclusion Criteria:

* sex worker living in the french antilles

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sex workers living in the french antilles
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge regarding HIV of Sex Workers in the French Antilles - Questionnaire Survey | one year
Attitudes regarding HIV of Sex Workers in the French Antilles - Questionnaire Survey | one year
Behaviours regarding HIV of Sex Workers in the French Antilles - Questionnaire Survey | one year
Practices regarding HIV of Sex Workers in the French Antilles - Questionnaire Survey | one year

IPD SHARING:
Plan to Share IPD: No